CLINICAL TRIAL: NCT03103581
Title: A Pilot Evaluation of BLI4700 Bowel Preparation in Adult Subjects
Brief Title: BLI4700-202: A Pilot Evaluation of BLI4700 Bowel Preparation in Adult Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Braintree Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLI4700-202
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-10

CONDITIONS: Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BLI4700 (Experimental): BLI4700 Bowel Preparation (Investigational Regimen)
  Interventions: Drug: BLI4700

INTERVENTIONS:
Drug: BLI4700 — BLI4700 Bowel Preparation (Investigational Regimen)

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of BLI4700 as a bowel preparation prior to colonoscopy in adult patients.

ELIGIBILITY:
Primary Inclusion Criteria:

1. Male or female outpatients who are undergoing colonoscopy for a routinely accepted indication.
2. At least 18 years of age
3. If female, and of child-bearing potential, is using an acceptable form of birth control.
4. Negative urine pregnancy test at screening, if applicable
5. In the Investigator's judgment, subject is mentally competent to provide informed consent to participate in the study

Primary Exclusion Criteria:

1. Subjects with known or suspected ileus, severe ulcerative colitis, gastrointestinal obstruction, gastric retention, bowel perforation, toxic colitis or megacolon.
2. Subjects who had previous significant gastrointestinal surgeries.
3. Subjects with uncontrolled pre-existing electrolyte abnormalities, or those with clinically significant electrolyte abnormalities based on Visit 1 laboratory results.
4. Subjects with a prior history of renal, liver or cardiac insufficiency
5. Subjects with impaired consciousness that predisposes them to pulmonary aspiration.
6. Subjects undergoing colonoscopy for foreign body removal and/or decompression.
7. Subjects who are pregnant or lactating, or intending to become pregnant during the study.
8. Subjects of childbearing potential who refuse a pregnancy test.
9. Subjects allergic to any preparation components.
10. Subjects who, in the opinion of the Investigator, should not be included in the study for any reason, including inability to follow study procedures.
11. Subjects who have participated in an investigational surgical, drug, or device study within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McGowan, MPH, Study Director — Braintree Laboratories, Inc.
Locations (2):
- United States (2):
  - Braintree Research Site 1, Anaheim, California
  - Braintree Research Site 2, Bastrop, Louisiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study protocol allowed for the evaluation of multiple formulations of BLI4700, however only a single formulation was evaluated in the trial. All data for that formulation is presented in a single arm.
Period: Overall Study
Arm/Group | BLI4700
Started | 17
Completed | 15
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: The study protocol allowed for the evaluation of multiple formulations of BLI4700, however only a single formulation was evaluated in the trial. All data for that formulation is presented in a single arm.
Arm/Group | BLI4700
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.9 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Successful Bowel Preparation
Description: Successful bowel preparation is defined as a preparation rated as Excellent or Good by the blinded endoscopist on a 4 point scale (Excellent, Good, Fair, Poor).
Time Frame: Day of colonoscopy
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | BLI4700
Number analyzed (Participants) | 17
Participants | 15

ADVERSE EVENTS:
Time Frame: 2 days
Description: The study protocol allowed for the evaluation of multiple formulations of BLI4700, however only a single formulation was evaluated in the trial. All data for that formulation is presented in a single arm.
Arm/Group | BLI4700
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 14/17
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BLI4700 (N=17)
abdominal distension (Gastrointestinal disorders) | 10
abdominal pain (Gastrointestinal disorders) | 1
abdominal pain upper (Gastrointestinal disorders) | 4
nausea (Gastrointestinal disorders) | 8
vomiting (Gastrointestinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sole disclosure restriction which sponsor imposes on the PI is a sixty (60) day limited restriction in order to the protect potentially proprietary information which may be patentable.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT03103581/Prot_SAP_000.pdf